CLINICAL TRIAL: NCT05779462
Title: Study of Pelvic Organ Mobility by Dynamic MRI in Pelvic Endometriosis
Brief Title: ENDOMETRIOSIS - MRI
Acronym: ENDO-MRI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0032; 2022-A02135-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis; Mobility Limitation; Magnetic Resonance Imaging; Diagnosis; Pelvis; Comparative Study
Keywords: Endometriosis ;; Mobility Limitation; Magnetic Resonance Imaging, Cine; Pelvis; Comparative Study
MeSH Terms: conditions — Endometriosis; Mobility Limitation; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with pelvic endometriosis: Patients referred for suspected pelvic endometriosis, with pelvic endometriosis on initial MRI
  Interventions: Other: Dynamic MRI Sequence
- patients without pelvic endometriosis: Patients referred for suspected pelvic endometriosis but without endometriosis found on diagnostic MRI.
  Interventions: Other: Dynamic MRI Sequence

INTERVENTIONS:
Other: Dynamic MRI Sequence — Addition of a Dynamic MRI Sequence during the MRI examination performed in routine care

SUMMARY:
Endometriosis is a frequent pathology with an estimated prevalence of 10% of women of childbearing age. There is no exact correspondence between the symptoms described by the patients and the severity of the lesions, which makes clinical diagnosis difficult. It therefore seems important to improve the complementary examinations available to make the diagnosis more precise and to better study the effectiveness of the treatments implemented. The clinical examination and per-surgical findings of patients with deep pelvic endometriosis show a clear decrease in the mobility of the pelvic organs in relation to each other, but few studies have looked at this mobility, which could however have an implication in explaining the pathophysiology of the disease and the symptomatology of the patients, as well as in the detection of lesions preoperatively. The persistence of hypo-mobility could also help to understand treatment failures.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for suspected pelvic endometriosis requiring pelvic MRI
* Female, nulliparous,
* patient with signed written consent, patient with health insurance,
* patient willing to comply with all study procedures and duration

Exclusion Criteria:

* BMI > 35,
* history of hereditary collagen and elastic tissue disease,
* history of pelviperitonitis,
* history of major pelvic surgery,
* inability to receive informed information,
* inability to participate in the entire study,
* lack of social security coverage,
* refusal to sign consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female, nulliparous
Study Population: The population concerns patients referred to the Lille University Hospital for suspected pelvic endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
the mean vertical displacement (in millimeters) measured on the anterior wall of the vagina between rest and maximum pushing force during dynamic MRI | Baseline

SECONDARY OUTCOMES:
the mean vertical displacement (in millimetres) measured on the cervix between rest and maximum thrust effort during dynamic MRI. | Baseline
the mean vertical displacement (in millimetres) measured on the posterior wall of the vagina between rest and maximum pushing force during dynamic MRI. | Baseline
the measurement of variation in mean vertical displacement (in millimetres) on the wall of each pelvic organ at the push effort between the initial dynamic MRI of patients with | Baseline
the statistical association between the symptoms of patients with endometriosis and the mean vertical displacement (in millimetres) on the wall of each pelvic organ at the push effort during dynamic MRI. | Baseline
  Initial symptoms are associated with initial dynamic MRI data and post therapeutic symptoms are associated with post-therapeutic dynamic MRI data.
  The symptoms of interest are dysmenorrhea, non-cyclic pelvic pain, dysuria, dychesia, transit disorders (diarrhea/constipation), and dyspareunia.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystele RUBOD, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service de chirurgie gynécologique Hôpital Jeanne de Flandre - CHU de LILLE, Lille, France